CLINICAL TRIAL: NCT05566236
Title: Study on the Effectiveness of an Evidence-based Board Game Project to Help Improve Tics and Interpersonal Interactions of Adolescents with Tourette Syndrome
Brief Title: Board Game Project for Adolescents with Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Chang Gung Children's Hospital (Other)
Responsible Party: Principal Investigator, Mei-Yin Lee, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201801998B0C501
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Tourette Syndrome in Adolescence; Social Adjustment; Psychosocial Functioning
Keywords: Tourette Syndrome; Depression; social adjustment; board game; Positive mental health
MeSH Terms: conditions — Social Adjustment; Tourette Syndrome; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- board game (Experimental): The participants received the usual standard of care(psychoeducation regarding Tourette Syndrome and one 50-mg tablet of pyridoxine daily), and they played the 60-minute parent-child board game at least once at home for consecutive 4 weeks.
  Interventions: Behavioral: board game
- Care as usual (No Intervention): The participants received the usual standard of care (psychoeducation regarding Tourette Syndrome and one 50-mg tablet of pyridoxine daily).

INTERVENTIONS:
Behavioral: board game — A board game was designed based on situated learning theory and the results of relevant studies. This board game contains a summary, answer booklet, and multiple card game tasks including situations of interpersonal interaction. The participants must discuss, share personal experiences, and find the answer together.
  Other Names: Non
  Arms: board game

SUMMARY:
The study aims to investigate the effectiveness of using a board game to improve adolescents' tics, mental health, and interpersonal interactions.

DETAILED DESCRIPTION:
This study utilizes a randomized control study design. According to the situated learning theory and qualitative research findings, this study develops a board game. This study enrolled adolescents with Tourette syndrome aged 12 to 18 as the subjects. Participants played board games at home at least once (about 60 minutes) a week for four consecutive weeks. The control group received the usual standard of care (psychoeducation regarding Tourette Syndrome and one 50-mg tablet of pyridoxine daily). The effectiveness indicators include self-reported status of positive mental health, tics severity, social adjustment, and depression by adolescents with TS.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 12 and 18 years were diagnosed with Tourette Syndrome or chronic tics disorder by a pediatrician, according to the DSM V.
* Ability to speak and understand Mandarin.
* Adolescents and their parents were willing to participate and fill in consent forms.

Exclusion Criteria:

· Adolescents with Tourette Syndrome have mental illness and serious diseases.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Positive Mental Health Scale | Pre-intervention (baseline), immediately after completion of the intervention (4 weeks after baseline) and at follow-up (12 weeks post-baseline).
  This study will use the Positive Mental Health Scale(25 items) to evaluate adolescents' degree of positive mental health. The lowest and highest total scores were 25 and 125, respectively. A high score indicates favorable positive mental health.
Yale Global Tic Severity Scale | Pre-intervention (baseline), immediately after completion of the intervention (4 weeks after baseline) and at follow-up (12 weeks post-baseline).
  The Yale Global Tic Severity Scale (YGTSS) will assess participants' motor and vocal tics' frequency, intensity, number, complexity, and interference. YGTSS also includes an overall Impairment Rating to determine each participant's interpersonal, academic, and occupational skill domains. Finally, the Global Severity Score will be acquired by adding the Total Motor Tic Score(0-25), Total Vocal Tic Score (0-25), and Overall Impairment Rating (0-50). The YGTSS has a total score ranging from 0 to 100, with the high score indicating a higher tics severity.

SECONDARY OUTCOMES:
Social adjustment scale for adolescents with Tourette syndrome | Pre-intervention (baseline), immediately after completion of the intervention (4 weeks after baseline) and at follow-up (12 weeks post-baseline).
  This study will use the social adjustment scale for adolescents with Tourette syndrome(17 items) to assess participants' level of social adjustment. The lowest and highest total scores were 17 and 68, respectively. A high score indicates favorable social adjustment.
Chinese Version Beck Youth Inventories II (depression inventory) | Pre-intervention (baseline), immediately after completion of the intervention (4 weeks after baseline) and at follow-up (12 weeks post-baseline).
  Chinese Version Beck Youth Inventories II (depression inventory)will used in this research to evaluate adolescents' depression. The depression inventory(20 items) has a total score ranging from 0 to 60, with a high score indicating a higher depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MY, Wang HS, Chen CJ, Lee MH. Social adjustment experiences of adolescents with Tourette syndrome. J Clin Nurs. 2019 Jan;28(1-2):279-288. doi: 10.1111/jocn.14564. Epub 2018 Jul 23. PMID 29893437
- [Background] Kennedy A, Semple L, Alderson K, Bouskill V, Karasevich J, Riske B, van Gunst S. Don't Push Your Luck! Educational Family Board (Not Bored) Game for School-Age Children Living with Chronic Conditions. J Pediatr Nurs. 2017 Jul-Aug;35:57-64. doi: 10.1016/j.pedn.2017.02.032. Epub 2017 Mar 14. PMID 28728770
- [Background] Malli MA, Forrester-Jones R, Murphy G. Stigma in youth with Tourette's syndrome: a systematic review and synthesis. Eur Child Adolesc Psychiatry. 2016 Feb;25(2):127-39. doi: 10.1007/s00787-015-0761-x. Epub 2015 Aug 28. PMID 26316059
- [Derived] Lee MY, Wang HS, Lien CY, Chen ZH. Effects of a Board Game on Tic Management and Psychosocial Functioning in Adolescents With Tourette Syndrome: Randomized Controlled Trial. JMIR Serious Games. 2025 Sep 9;13:e76208. doi: 10.2196/76208. PMID 40925588